CLINICAL TRIAL: NCT01463657
Title: A Phase 2 Bilateral (Split-face) Comparison Study to Assess Two Formulations of ELAPR Compared to Juvéderm® Ultra Plus for the Treatment of Moderate to Severe Nasolabial Folds
Brief Title: Split-face Comparison Study to Assess ELAPR Compared to Juvéderm® for the Treatment of Nasolabial Folds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elastagen Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ELAPR P2
Record Dates: First submitted 2011-09-18; First posted 2011-11-02 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Aging
Keywords: Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELAPR002 (Experimental): Each treatment will consist of up 15 injections in total, each consisting of up to 0.1 ml of product, delivered to the mid to deep dermis of the skin of each NLF using a 27G needle. The needle will be inserted at an approximate angle of 30o parallel to the skin, and the product may be injected by a retrograde injection or by deposition of a bolus. ELAPR and the control may be implanted parallel or perpendicular to the NLF. Exactly the same technique will be used for the treatment of both NLFs for each patient.
  Interventions: Device: ELAPR002
- Juvéderm® Ultra Plus (Active Comparator): Each treatment will consist of up 15 injections in total, each consisting of up to 0.1 ml of product, delivered to the mid to deep dermis of the skin of each NLF using a 27G needle. The needle will be inserted at an approximate angle of 30o parallel to the skin, and the product may be injected by a retrograde injection or by deposition of a bolus. ELAPR and the control may be implanted parallel or perpendicular to the NLF. Exactly the same technique will be used for the treatment of both NLFs for each patient.
  Interventions: Device: Juvéderm® Ultra Plus

INTERVENTIONS:
Device: Juvéderm® Ultra Plus — Patients will receive either ELAPR002b or ELAPR002d for the treatment of one NLF, and Juvéderm® Ultra Plus for the treatment of the second, opposite NLF. Treatments will be provided on Day 1 and repeated on Day 29 (if required at the discretion of the investigator) Day 57 (if required at the discretion of the investigator)to achieve OCR.
  Arms: Juvéderm® Ultra Plus
Device: ELAPR002 — Each treatment will consist of up 15 injections in total, each consisting of up to 0.1 ml of product, delivered to the mid to deep dermis of the skin of each NLF using a 27G needle. The needle will be inserted at an approximate angle of 30o parallel to the skin, and the product may be injected by a retrograde injection or by deposition of a bolus. ELAPR and the control may be implanted parallel or perpendicular to the NLF. Exactly the same technique will be used for the treatment of both NLFs for each patient.
  Other Names: Tropelastin
  Arms: ELAPR002

SUMMARY:
Patients presenting to the clinic for treatment of moderate to severe Nasolabial folds will be recruited to receive either ELAPR002b or ELAPR002d for the treatment of one Nasolabial fold and Juvéderm® Ultra Plus for the treatment of the second, opposite Nasolabial fold.

DETAILED DESCRIPTION:
The treatment will be repeated on Day 29 (if required) and Day 57 (if required) to achieve optimum cosmetic results (OCR).

Each treatment will consist of up to 15 injections in total, each consisting of up to 0.1 ml of product, delivered to the mid to deep dermis of the skin of each Nasolabial fold using a 27G needle.

Each patient will receive the same preparation implanted as a bolus of 0.1mL at Day 1 into the mid-deep dermis of the skin of the medial aspect of the upper arm using a 27G needle, and two 2mm biopsies will be taken at the same visit on Day 57, Day 85 or Day 169 depending on randomisation for histopathology assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 - 65 years
* Male or Female
* Moderate to severe NLFs scored equally as a 3 or 4 out of 5 on both sides of the face using the WAS scale
* Good general health status
* Able to give informed consent

Exclusion Criteria:

* Clinically significant abnormalities of haematology or biochemistry testing
* Bleeding diathesis, anticoagulant drugs, thrombocytopenia or clinically significant prolonged bleeding time
* Chronic use of aspirin, other non-steroidal anti-inflammatory drugs or other anti-platelet agents
* Allergy to local anaesthetics
* Active infection at the treatment site
* Treatment of either NLF other than with a hyaluronic acid (HA) dermal filler and treatment with a HA dermal filler within 18 months of enrolment
* Any serious medical condition which in the opinion of the investigator would have a strong possibility of requiring systemic corticosteroid medication
* Pregnancy/lactation
* History of keloid formation
* Systemic corticosteroids within last 12 weeks
* Diabetes or metabolic disorders
* A history of anaphylaxis or allergic reactions including any known hypersensitivity to Hyaluronic acid or lidocaine
* Sensitivity to Juvéderm® Ultra Plus or Juvéderm® products.
* Participation in any other clinical trial one month prior to treatment and for the duration of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assess the effect of two formulations of ELAPR on change from baseline of the severity of the Nasolabial folds against a Wrinkle Assessment Scale of Nasolabial folds score at 24 weeks vs. active control | 24 weeks
  The primary efficacy variable is the change in Wrinkle Assessment Scale (WAS). The values for WAS recorded at each visit will be summarized by treatment.

SECONDARY OUTCOMES:
Assess the acute safety of ELAPR | 24 weeks
  Adverse event profile will be collected.
Assess chronic safety of ELAPR | 24 weeks
  A serum sample will be collected at Day 1, 29, 85, and Day 169, or at the completion visit in the event of early withdrawal or early termination and stored for a maximum of 5 years for the development of an assay to measure circulating anti-tropoelastin antibody levels.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Goodman, MBBS FRACS, Principal Investigator — Dermatology Institute of Victoria
Locations (2):
- Australia (2):
  - Cosmedic, Southport, Queensland
  - Dermatology Institute of Victoria, Melbourne, Victoria